CLINICAL TRIAL: NCT03881111
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial of Pembrolizumab (MK-3475) in Combination With Cisplatin and 5-Fluorouracil Versus Placebo in Combination With Cisplatin and 5-Fluorouracil as First-Line Treatment in Subjects With Advanced/Metastatic Esophageal Carcinoma (KEYNOTE-590)
Brief Title: First-line Esophageal Carcinoma Study With Chemo vs. Chemo Plus Pembrolizumab (MK-3475-590/KEYNOTE-590)-China Extension Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to protocol amendment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-590 China Extension; 2017-000958-19 (EudraCT Number); 173739 (Registry Identifier: JAPIC-CTI); MK-3475-590 (Other: Merck Protocol Number); KEYNOTE-590 (Other: Merck)
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Neoplasms
Keywords: Programmed Cell Death-1 (PD-1); Programmed Cell Death 1 (PD1); Programmed Cell Death-Ligand 1 (PD-L1, PDL1); Programmed Cell Death-Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Esophageal Neoplasms | interventions — pembrolizumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Cisplatin + 5-FU (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W), cisplatin 80 mg/m^2 IV Q3W, and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours). All treatments will be administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: 5-FU
- Placebo + Cisplatin + 5-FU (Placebo Comparator): Participants receive placebo to pembrolizumab (saline) IV Q3W, cisplatin 80 mg/m^2 IV Q3W, and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours). All treatments will be administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: 5-FU

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg administered IV Q3W on Day 1 of each 3-week cycle, up to 35 administrations.
  Other Names: MK-3475
  Arms: Pembrolizumab + Cisplatin + 5-FU
Drug: Placebo — Placebo to pembrolizumab (saline) administered IV Q3W on Day 1 of each 3-week cycle, up to 35 administrations.
  Arms: Placebo + Cisplatin + 5-FU
Drug: Cisplatin — 80 mg/m^2 administered IV Q3W on Day 1 of each 3-week cycle. Duration of cisplatin treatment will be capped at 6 doses.
Drug: 5-FU — 800 mg/m^2/day (4000 mg/m^2 total per cycle) administered as continuous IV infusion on Days 1 to 5 (120 hours) of each 3-week cycle, or per local standard for 5-FU administration.

SUMMARY:
The purpose of this Chinese extension study is to evaluate efficacy and safety of pembrolizumab plus cisplatin and 5-fluorouracil (5-FU) chemotherapy versus placebo plus cisplatin and 5-FU chemotherapy as first-line treatment in a Chinese cohort of participants with locally advanced or metastatic esophageal carcinoma.

The primary efficacy hypotheses are that both progression-free survival (PFS), according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and determined by blinded independent central review, and overall survival (OS) are superior with pembrolizumab plus chemotherapy compared with placebo plus chemotherapy in all Chinese participants as well as Chinese participants whose tumors are programmed cell death-ligand 1 (PD-L1)-positive.

DETAILED DESCRIPTION:
The Chinese extension to MK-3475-590 (NCT03189719) will enroll a total of approximately 90 participants.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the esophagogastric junction (EGJ)
* Has measurable disease per RECIST 1.1 as determined by the local site investigator/radiology assessment
* Eastern Cooperative Group (ECOG) performance status of 0 to 1
* Can provide either a newly obtained or archival tissue sample for PD-L1 by immunohistochemistry analysis
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to randomization and be willing to use an adequate method of contraception (e.g. abstinence, intrauterine device, diaphragm with spermicide, etc.) for the course of the study through 120 days after the last dose of study treatment and up to 180 days after last dose of cisplatin
* Male participants of childbearing potential must agree to use an adequate method of contraception (e.g. abstinence, vasectomy, male condom, etc.) starting with the first dose of study treatment through 120 days after the last dose of study treatment and up to 180 days after last dose of cisplatin, and refrain from donating sperm during this period
* Has adequate organ function

Exclusion Criteria:

* Has locally advanced esophageal carcinoma that is resectable or potentially curable with radiation therapy (as determined by local investigator)
* Has had previous therapy for advanced/metastatic adenocarcinoma or squamous cell cancer of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the EGJ
* Has had major surgery, open biopsy, or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study treatment
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early-stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, in situ breast cancer that has undergone potentially curative therapy, and in situ or intramucosal pharyngeal cancer
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment, or has a history of organ transplant, including allogeneic stem cell transplant
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis, or has an active infection requiring systemic therapy
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study medication and up to 180 days after last dose of cisplatin
* Has received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor or has previously participated in a pembrolizumab (MK-3475) clinical trial
* Has severe hypersensitivity (≥ Grade 3) to any study treatment (pembrolizumab, cisplatin, or 5-FU) and/or any of its excipients
* Has a known history of active tuberculosis (TB; Mycobacterium tuberculosis) or human immunodeficiency virus (HIV) infection
* Has known history of or is positive for hepatitis B or hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Has had radiotherapy within 14 days of randomization. Participants who received radiotherapy >14 days prior to randomization must have completely recovered from any radiotherapy-related AEs/toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-05-11 (Estimated); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in all participants | Up to 2 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first. For this analysis, PFS will be assessed in all participants.
PFS per RECIST Version 1.1 in PD-L1 biomarker-positive participants | Up to 2 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first. For this analysis, PFS will be assessed in PD-L1 biomarker-positive participants.
Overall Survival (OS) in all participants | Up to 2 years
  OS is defined as the time from randomization to death due to any cause. For this analysis, OS will be assessed in all participants.
OS in PD-L1 biomarker-positive participants | Up to 2 years
  OS is defined as the time from randomization to death due to any cause. For this analysis, OS will be assessed in PD-L1 biomarker-positive participants.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 in all participants | Up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this analysis, ORR will be assessed in all participants.
ORR per RECIST 1.1 in PD-L1 biomarker-positive participants | Up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this analysis, ORR will be assessed in PD-L1 biomarker-positive participants.
Duration of Response (DOR) per RECIST 1.1 in all participants | Up to 2 years
  For participants who demonstrate CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), DOR is defined as the time from first documented evidence of CR or PR until disease progression per RECIST 1.1 based on assessments by blinded independent central review or death due to any cause, whichever occurs first. For this analysis, DOR will be assessed in all participants.
DOR per RECIST 1.1 in PD-L1 biomarker-positive participants | Up to 2 years
  For participants who demonstrate CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), DOR is defined as the time from first documented evidence of CR or PR until disease progression per RECIST 1.1 based on assessments by blinded independent central review or death due to any cause, whichever occurs first. For this analysis, DOR will be assessed in PD-L1 biomarker-positive participants.
Number of participants with an adverse event (AE) | Up to 27 months
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Number of participants discontinuing study treatment due to an AE | Up to 2 years
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Change from baseline in the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) Score | Baseline, End of Treatment (~1 year)
  The EORTC QLQ-C30 was developed to assess the quality of life of patients with cancer. It contains 30 questions (items), 24 of which aggregate into nine multi-item scales representing various aspects, or dimensions, of quality of life (QOL): one global scale, five functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea, pain), and six additional single-symptom items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease. Individual items are scored on a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Raw scores for each scale are standardized into a range of 0 to 100 by linear transformation; a higher score on the global and functional scales represents a higher ("better") level of functioning, and a higher score on the symptom scale represents a higher ("worse") level of symptoms.
Change from baseline in the EORTC Quality Of Life Questionnaire Oesophageal Module (QLQ-OES18) Score | Baseline, End of Treatment (~1 year)
  The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer. It contains 18 items and is based on four subscales-dysphagia (three items), eating (four items), reflux (two items) and pain (three items), as well as six single-item subscales-saliva swallowing, choking, dry mouth, taste, cough and speech. All items are scored using a four-point Likert scale that offers these response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores are standardized into a range of 0 to 100 by linear transformation; higher symptom scores represent a higher ("worse") level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (20):
- China (20):
  - Anhui Provincial Hospital ( Site 0106), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University ( Site 0112), Hefei, Anhui
  - Peking Union Medical College Hospital ( Site 0123), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 0119), Xiamen, Fujian
  - Guangdong General Hospital ( Site 0103), Guangzhou, Guangdong
  - The Affiliated Tumour Hospital of Harbin Medical University ( Site 0102), Harbin, Heilongjiang
  - Hunan Cancer Hospital ( Site 0105), Changsha, Hunan
  - PLA Cancer Centre of Nanjing Bayi Hospital ( Site 0110), Nanjing, Jiangsu
  - Jiangsu Cancer Hospital ( Site 0117), Nanjing, Jiangsu
  - Zhongda Hospital Southeast University ( Site 0125), Nanjing, Jiangsu
  - Jilin Cancer Hospital ( Site 0101), Changchun, Jilin
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0120), Xi'an, Shannxi
  - Zhejiang Cancer Hospital ( Site 0116), Hangzhou, Zhejiang
  - Beijing Cancer Hospital ( Site 0100), Beijing
  - Fujian Provincial Cancer Hospital ( Site 0104), Fuzhou
  - Shanghai Chest Hospital ( Site 0111), Shanghai
  - Fudan University Shanghai Cancer Center ( Site 0108), Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0114), Shanghai
  - Tongji Medical College Huazhong University of Science and Technology ( Site 0109), Wuhan
  - Henan Cancer Hospital ( Site 0107), Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php